CLINICAL TRIAL: NCT05970640
Title: Phase Ib Trial to Assess Safety and Tolerability of Multiple Subcutaneous Doses of BI 3006337 in Patients With Overweight or Obesity and Hepatic Steatosis
Brief Title: A Study to Test How Well Different Doses of BI 3006337 Are Tolerated by People With Overweight or Obesity and With Fatty Liver Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1466-0002
Record Dates: First submitted 2023-07-21; First posted 2023-08-01 (Actual); Results first posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Non-alcoholic Fatty Liver Disease; Obesity
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BI 3006337 50 mg (Experimental): Subject with overweight/obesity and steatosis received subcutaneous solution for administration of 50 milligram of BI 3006337 once weekly.
  Interventions: Drug: BI 3006337
- BI 3006337 100 mg (Experimental): Subjects with overweight/obesity and steatosis received subcutaneous solution for administration of 100 milligram of BI 3006337 once weekly.
  Interventions: Drug: BI 3006337
- BI 3006337 150 mg (Experimental): Subjects with overweight/obesity and steatosis received subcutaneous solution for administration of 150 milligram of BI 3006337 once weekly.
  Interventions: Drug: BI 3006337
- Placebo (Placebo Comparator): Subjects with overweight/obesity and steatosis received subcutaneous solution for administration of Placebo once weekly.
  Interventions: Drug: Placebo matching BI 3006337

INTERVENTIONS:
Drug: BI 3006337 — Subject with overweight/obesity and steatosis received subcutaneous solution once weekly.
  Arms: BI 3006337 100 mg; BI 3006337 150 mg; BI 3006337 50 mg
Drug: Placebo matching BI 3006337 — Subject with overweight/obesity and steatosis received subcutaneous solution once weekly.
  Arms: Placebo

SUMMARY:
This study is open to adults with overweight or obesity who also have fatty liver disease. The purpose of this study is to find the highest dose of BI 3006337 that people with overweight or obesity and with fatty liver disease can tolerate.

Participants are divided into 4 groups of equal size randomly, which means by chance. Different doses of BI 3006337 are given to participants in each group. Participants in each group receive an injection of either BI 3006337 or placebo once a week. Placebo injections look like BI 3006337 injections but do not contain any medicine.

Participants are in the study for about 4 months. During this time, they visit the study site 18 times. Three of the visits include overnight stays at the study site. The doctors check the health of the participants and note any health problems that could have been caused by BI 3006337.

ELIGIBILITY:
Inclusion Criteria:

- Male or female trial participants ≥18 years and ≤75 years of age at time of consent.

Women of child-bearing potential (WOCBP) must be willing and able to use 2 forms of effective contraception where at least 1 form is a highly effective method of birth control per ICH M3 (R2) that results in a low failure rate of less than 1% per year when used consistently and correctly. Male trial participants must be willing and able to use condom if their partner is a WOCBP

* Body mass index (BMI) ≥25 - <40 kg/m^2
* Liver fat fraction ≥8% as measured by Magnetic resonance imaging proton density fat fraction (MRI-PDFF)
* Signed and dated written informed consent in accordance with International Council for Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial

Exclusion Criteria:

- Current or past significant alcohol consumption (daily alcohol consumption in women should not exceed more than one standard drink per day and two drinks per day for men, whereby one standard drink is equivalent to 12 oz beer [5% alcohol]; 5 ounces of wine [12% alcohol], 1.5 ounces of 80 proof [40% alcohol]) or inability to reliably quantify alcohol consumption based on Investigator judgement within the last 5 years.

The Alcohol Use Disorders Identification Test (AUDIT) shall be used a standardized screening tool for alcohol use disorder

* Intake of medications historically associated with liver injury, hepatic steatosis, or steatohepatitis (e.g. oral or intravenous corticosteroids, methotrexate, valproic acid, tamoxifen, tetracycline, amiodarone) for more than 14 consecutive days within 12 weeks prior to the screening visit
* Presence of any form of acute or chronic liver disease other than simple steatosis (e.g. viral hepatitis, autoimmune liver disease, primary biliary sclerosis, primary sclerosing cholangitis, Wilson's disease, hemochromatosis, alpha-1 antitrypsin deficiency). Chronic viral hepatitis parameters that would be considered exclusionary for the participation to this trial are (hepatitis B and C testing will be done at the screening visit):

  * Hepatitis B virus (HBV): trial participants with positive Hepatitis B virus surface antigen (HbsAg)
  * Hepatitis C virus (HCV): trial participants with positive HCV RNA. Trial participants treated for hepatitis C must have a negative RNA test at screening and also be HCV RNA negative for at least 3 years prior to screening in order to be eligible for the trial
* Liver stiffness >10 Kilopascal (kPa) as measured using Fibroscan. In patients with a non-valid Fibroscan measurement, a Fib-4 score >1.3 should be considered exclusionary.
* Suspicion, confirmed diagnosis, or history of hepatocellular carcinoma
* Treatment with vitamin E (at a minimum dose of 800 IU/day) or pioglitazone not stable (in the opinion of the Investigator) within 90 days before screening
* History of type 1 diabetes
* Use of Glucagon-like peptide 1 (GLP1)-receptor agonists within last 90 days before screening Further exclusion criteria apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-08-14 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-11-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Velocity Clinical Research-Chula Vista, Chula Vista, California
  - Velocity Clinical Research-La Mesa-69117, La Mesa, California
  - Catalina Research Institute, LLC-Montclair-49051, Montclair, California
  - Accel Research Sites-Deland-67606, DeLand, Florida
  - Floridian Clinical Research-Miami Lakes-68368, Miami Lakes, Florida
  - iResearch Atlanta, Decatur, Georgia
  - Centricity Research-Columbus-68879, Columbus, Ohio
  - AMR Knoxville, Knoxville, Tennessee
  - The Liver Institute at Methodist Dallas, Dallas, Texas
  - American Research Corporation at the Texas Liver Institute, San Antonio, Texas
  - Endeavor Clinical Trials, San Antonio, Texas
  - Velocity Clinical Research-West Jordan-69043, West Jordan, Utah

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was single-blind and randomised trial with placebo matching the dose of BI 3006337 as comparator. Treatment allocation was performed within each dose group in a 5:2 ratio (BI 3006337 to placebo). Participants were included in the trial once they had signed the informed consent. The trial consisted of a screening period of up to 6 weeks to assess participant eligibility, a treatment period of 12 weeks and a follow-up period of 3 weeks.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated. Of 64 enrolled, 63 began treatment; one participant in the BI 3006337 150 mg group withdrew consent before Day -1 and underwent no procedures.
Period: Overall Study
Arm/Group | BI 3006337 50 mg | BI 3006337 100 mg | BI 3006337 150 mg | Placebo
Started | 11 | 10 | 23 | 19
Completed | 10 | 7 | 20 | 17
Not Completed | 1 | 3 | 3 | 2
Not completed — Adverse Event | 1 | 3 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1
Not completed — Sponsor decision | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Treated set (TS): TS includes all subjects from the randomised set who are treated with at least one dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 3006337 50 mg | BI 3006337 100 mg | BI 3006337 150 mg | Placebo | Total
Number analyzed (Participants) | 11 | 10 | 23 | 19 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (9.3) | 45.5 (16.1) | 54.4 (11.9) | 51.5 (14.0) | 50.0 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 9 | 10 | 26
  Male | 8 | 6 | 14 | 9 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 7 | 22 | 15 | 52
  Not Hispanic or Latino | 3 | 3 | 1 | 4 | 11
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 11 | 8 | 23 | 17 | 59
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 0 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Drug-related Adverse Events (AEs)
Description: Number of subjects with drug-related adverse events (AEs) occurring between first administration of trial medication (BI 3006337 or placebo) and end of study (EOS) is reported.
Time Frame: From drug administration of BI 3006337 until end of the treatment, up to 99 days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- BI 3006337 50 mg: Subjects with overweight/obesity and steatosis received subcutaneous solution for administration of 50 milligram of BI 3006337 once weekly.
Arm/Group | BI 3006337 50 mg | BI 3006337 100 mg | BI 3006337 150 mg | Placebo
Number analyzed (Participants) | 11 | 10 | 23 | 19
Participants | 9 | 8 | 14 | 5

2. Secondary Outcome: Area Under the Concentration-time Curve of BI 3006337 in Serum Over the Dosing Interval Tau at Steady State (AUCτ,ss) After the Last Dose in Week 12
Description: Area under the concentration-time curve of BI 3006337 in serum over the dosing interval tau at steady state (AUCτ,ss) after the last dose in Week 12 is reported.
Time Frame: 0 hours (prior to drug administration) and 3, 7, 11, 15, 23, 27, 31, 35, 39, 47, 72, 168 and 504 hours after drug administration in week 12
Population: Pharmacokinetic parameter analysis set (PKS): This set includes all trial participants in the treated set (TS) who provide at least one primary or secondary PK endpoint that was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability. One subject from the 50 mg arm was excluded from the analysis due to a missing sample, which precluded characterization of the elimination phase.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*Microgram/Liter
Groups:
- BI 3006337 100 mg: Subject with overweight/obesity and steatosis received subcutaneous solution for administration of 100 milligram of BI 3006337 once weekly.
- BI 3006337 150 mg: Subject with overweight/obesity and steatosis received subcutaneous solution for administration of 150 milligram of BI 3006337 once weekly.
Arm/Group | BI 3006337 50 mg | BI 3006337 100 mg | BI 3006337 150 mg
Number analyzed (Participants) | 9 | 7 | 19
Hour*Microgram/Liter | 21000 (57.3) | 38800 (81.1) | 67100 (50.4)

3. Secondary Outcome: Maximum Measured Concentration of BI 3006337 in Serum at Steady State (Cmax,ss) After the Last Dose in Week 12
Description: Maximum measured concentration of BI 3006337 in serum at steady state (Cmax,ss) after the last dose in Week 12 is reported.
Time Frame: 0 hours (prior to drug administration) and 3, 7, 11, 15, 23, 27, 31, 35, 39, 47, 72, 168 hours after drug administration in week 12
Population: Pharmacokinetic parameter analysis set (PKS): This set includes all trial participants in the treated set (TS) who provide at least one primary or secondary PK endpoint that was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram/Liter
Arm/Group | BI 3006337 50 mg | BI 3006337 100 mg | BI 3006337 150 mg
Number analyzed (Participants) | 10 | 7 | 19
Microgram/Liter | 312 (87.7) | 761 (64.9) | 1060 (64.2)

4. Secondary Outcome: Time From Dosing to the Maximum Measured Concentration of BI 3006337 in Serum at Steady State (Tmax,ss) After the Last Dose in Week 12
Description: Time from dosing to the maximum measured concentration of BI 3006337 in serum at steady state (tmax,ss) after the last dose in Week 12 is reported.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Median (Full Range); unit: Hour
Arm/Group | BI 3006337 50 mg | BI 3006337 100 mg | BI 3006337 150 mg
Number analyzed (Participants) | 10 | 7 | 19
Hour | 13 [11 to 47] | 15 [3 to 35] | 27 [7 to 47]

5. Secondary Outcome: Relative Percentage Change in Liver Steatosis From Baseline After 12 Weeks of Treatment
Description: Relative percentage change in liver steatosis from baseline after 12 weeks of treatment is reported. Liver steatosis is measured by Magnetic resonance imaging proton density fat fraction (MRI-PDFF).
Time Frame: Baseline (-48 to -4): the last observed measurement prior to drug administration, Day 85
Population: Treated set (TS): The TS includes all subjects from the randomised set who are treated with at least one dose of study medication. The treatment assignment will be determined based on the first treatment the trial subjects received. The TS is the basis for safety analyses. The main efficacy analysis was conducted using the Treated Set and excluded all participants who discontinued due to Coronavirus disease 2019 (COVID-19). Only subjects with available data at baseline and week 12 were included.
Measure: Mean (Standard Deviation); unit: Percent change
Groups:
- Placebo: Subject with overweight/obesity and steatosis received subcutaneous solution for administration of Placebo once weekly.
Arm/Group | BI 3006337 50 mg | BI 3006337 100 mg | BI 3006337 150 mg | Placebo
Number analyzed (Participants) | 10 | 10 | 22 | 18
Percent change | -13.01 (21.92) | -16.59 (40.28) | -39.21 (14.73) | 6.13 (35.24)

ADVERSE EVENTS:
Time Frame: From drug administration of BI 3006337 until end of the treatment, up to 99 days
Description: Treated set (TS): TS includes all subjects from the randomised set who are treated with at least one dose of study medication.
Arm/Group | BI 3006337 50 mg | BI 3006337 100 mg | BI 3006337 150 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10 | 0/23 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10 | 1/23 | 0/19
Other Adverse Events (participants affected / at risk) | 10/11 | 9/10 | 18/23 | 15/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BI 3006337 50 mg (N=11) | BI 3006337 100 mg (N=10) | BI 3006337 150 mg (N=23) | Placebo (N=19)
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 3006337 50 mg (N=11) | BI 3006337 100 mg (N=10) | BI 3006337 150 mg (N=23) | Placebo (N=19)
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Middle ear effusion (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 2 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal wall pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 2 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 2 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 4 | 1
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Faeces soft (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 4 | 2 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2 | 1 | 1
Chest discomfort (General disorders) | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 0 | 1
Injection site erythema (General disorders) | 3 | 3 | 2 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 1
Injection site pruritus (General disorders) | 2 | 0 | 2 | 0
Injection site reaction (General disorders) | 3 | 5 | 6 | 0
Vessel puncture site haematoma (General disorders) | 0 | 0 | 0 | 1
Vessel puncture site pain (General disorders) | 0 | 0 | 0 | 2
Sunscreen sensitivity (Immune system disorders) | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 1 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 1 | 3
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 2
Viral infection (Infections and infestations) | 1 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 2 | 0
Lipase increased (Investigations) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 4 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 4 | 0
Hyperphagia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 4 | 1 | 2 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Myalgia intercostal (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 3 | 2 | 5 | 4
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 2 | 0 | 0 | 0
Libido decreased (Psychiatric disorders) | 0 | 1 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Crystalluria (Renal and urinary disorders) | 1 | 1 | 3 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urine odour abnormal (Renal and urinary disorders) | 0 | 0 | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2024-02-08): https://cdn.clinicaltrials.gov/large-docs/40/NCT05970640/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-28): https://cdn.clinicaltrials.gov/large-docs/40/NCT05970640/SAP_001.pdf